CLINICAL TRIAL: NCT00000669
Title: A Phase I Safety and Pharmacokinetics Study of 2',3'-Dideoxyinosine (ddI) Administered Twice Daily to Infants and Children With AIDS or Symptomatic HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 091; 070V1; AI454-003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 1996-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
To determine the safety and maximum tolerated dose (MTD) of 2',3'-dideoxyinosine (ddI), given orally and intravenously, in infants and children with AIDS. The study also measures bloodstream and cerebrospinal fluid (CSF) levels of the administered drug, and provides a preliminary assessment of the effectiveness of ddI on HIV replication.

AMENDED: Based on safety established in the first dosing phase of 52 weeks and long term dosing data in adults, the dosing period will be extended to 104 weeks. Original design: Information presently available indicates that ddI has high antiviral activity with less apparent toxicity than zidovudine (AZT) (the drug presently used to treat AIDS).

DETAILED DESCRIPTION:
AMENDED: Based on safety established in the first dosing phase of 52 weeks and long term dosing data in adults, the dosing period will be extended to 104 weeks. Original design: Information presently available indicates that ddI has high antiviral activity with less apparent toxicity than zidovudine (AZT) (the drug presently used to treat AIDS).

AMENDED: Dosing will proceed for 104 weeks at each dose level. Original design: Five patients are treated at the initial dose level. Because ddI is not stable in the acid environment of the stomach, oral doses of ddI follow administration of an antacid. An alternative method of dosing is to mix the reconstituted ddI with an appropriate volume of Maalox TC or Mylanta II. In order to determine the MTD, successive groups of 5 patients enter the study at a higher dose level after 3 patients have experienced 3 weeks of dosing and significant toxicities have not developed. Patients are assigned to treatment groups in the order in which they are enrolled. Dosing proceeds for 16 weeks at each dose level. However, consideration is given to escalating patients entered at the lowest dose to the next dose level after 10 weeks of dosing. The dose escalation continues until toxicities requiring dose modifications are found in 2 of 5 in any group.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis if this drug is extended to children.
* Acute therapy not exceeding 7 days with oral or intravenous acyclovir for herpes simplex infections.
* Trimethoprim / sulfamethoxazole for Pneumocystis carinii infections during course of study at discretion of investigator after discussion with the sponsor.
* Symptomatic therapy with analgesics, antihistamines, antiemetics, antidiarrheal agents, or other supportive therapy as deemed necessary by the principal investigator.

Patients must have:

* Diagnosis of AIDS as defined by CDC or meeting CDC P2 classification.
* Patients must be free of opportunistic infection or other serious bacterial, fungal, or parasitic infection at time of entry into study.
* Life expectancy > 6 months.
* Parent or guardian (and patient as applicable) able to give informed consent.
* Available for follow-up for at least 6 months.
* Allowed: Hemophilia.

Exclusion Criteria

Co-existing Condition:

Children with the following are excluded:

* Chronic hematologic disorders unrelated to coagulation defects, hemoglobinopathies, or ITP.
* Intractable diarrhea.
* No venous access.
* History of seizures within previous 2 years or currently requiring anticonvulsants for control.
* Currently active heart disease as evidenced by a cardiac arrhythmia or other significant abnormality on routine electrocardiography (ECG) or shortening fraction of < 10 percent on echocardiogram.
* Renal disease.
* Any other clinical condition that in the opinion of the investigator makes the patient unsuitable for study.

Concurrent Medication:

Excluded:

* Antiretroviral drugs.
* Zidovudine (AZT).
* AL 721.
* Interferon.
* Corticosteroids.
* Immunomodulating drugs.
* Other systemic investigation agent.
* Ribavirin.
* Rifampin, barbiturates, or any other potent inducer or inhibitor of drug-metabolizing enzymes.
* Cytotoxic anticancer therapy.
* H-2 blockers.
* Intravenous ketoconazole.
* Immunoglobulin preparations.

Children with the following are excluded:

* Chronic hematologic disorders unrelated to coagulation defects, hemoglobinopathies, or ITP.
* Intractable diarrhea.
* No venous access.
* History of seizures within previous 2 years or currently requiring anticonvulsants for control.
* Currently active heart disease as evidenced by a cardiac arrhythmia or other significant abnormality on routine electrocardiography (ECG) or shortening fraction of < 10 percent on echocardiogram.
* Renal disease.
* Any other clinical condition that in the opinion of the investigator makes the patient unsuitable for study.
* Renal disease.

Prior Medication:

Excluded:

* Any prior therapy which in the opinion of the investigator would make the patient unsuitable for study.

Excluded within 2 weeks of study entry:

* Trimethoprim / sulfamethoxazole.

Excluded within 1 month of study entry:

* Study drug or other antiretroviral drug or systemic investigational agent.
* Any agent known as a potent inducer or inhibitor of drug metabolizing enzymes.
* H-2 blockers.
* Ketoconazole.
* Immunoglobulin preparations.

Excluded within 3 months of study entry:

* Ribavirin.

Excluded:

* Zidovudine (AZT) for > 6 months.
* Cytotoxic anticancer therapy.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Blood transfusion.
* Lymphocyte transfusions for immune reconstitution.
* Bone marrow transplant.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25

CONTACTS AND LOCATIONS:
Overall Officials: Scott GB, Study Chair
Locations (5):
- United States (5):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Miami School of Medicine, Miami, Florida
  - The Regional Medical Ctr, Memphis, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas

REFERENCES:
- [Background] Butler KM, Husson RN, Balis FM, Brouwers P, Eddy J, el-Amin D, Gress J, Hawkins M, Jarosinski P, Moss H, et al. Dideoxyinosine in children with symptomatic human immunodeficiency virus infection. N Engl J Med. 1991 Jan 17;324(3):137-44. doi: 10.1056/NEJM199101173240301. PMID 1670591